CLINICAL TRIAL: NCT07256535
Title: Blood Bupivacaine Concentration After Transversus Abdominis Plane Block and Quadratus Lumborum Block in Pediatric Patients: A Randomized Controlled Trial
Brief Title: Blood Bupivacaine Concentration After Regional Block Applications in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KAEK/18.bI.07
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Blood Bupivacaine Concentration
Keywords: Pediatric Population; Transversus Abdominis Plan Block; Quadratus Lumborum Block; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP USING Transversus Abdominis Plane Block (Active Comparator): After induction of general anesthesia in all patients, once airway security is ensured, the standard regional anesthesia technique will be performed under ultrasound guidance by the same physician. A transversus abdominis plane block will be performed using an in-plane approach, passing through the external oblique and internal oblique muscles visible on ultrasound, and then advancing toward the fascial layer separating the internal oblique and transversus abdominis muscles. Following the block, the surgical team will begin the procedure. Thirty and sixty minutes after the block, 2 mL of blood will be collected into a routine biochemistry tube, and the blood bupivacaine level will be measured.
  Interventions: Procedure: Transversus Abdominis Plane Block
- GROUP USING Quadratus Lumborum Block (Active Comparator): After induction of general anesthesia in all patients, once airway security is ensured, the standard regional anesthesia technique will be performed by the same person under ultrasound guidance. The ultrasound probe is placed transversely, just above the iliac crest in the midaxillary line. After visualizing the vertebral body, transverse process, psoas major, quadratus lumborum, and erector spinae muscles, a local anesthetic will be administered between the quadratus lumborum and psoas major muscles, using an in-plane approach, as visible on ultrasound. Thirty and 60 minutes after the block, 2 mL of blood will be collected in a routine biochemistry tube, and the blood bupivacaine level will be measured.
  Interventions: Procedure: Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block — transversus abdominis plane block will be performed using 0.25-0.5% cc/kg bupivacaine
  Arms: GROUP USING Transversus Abdominis Plane Block
Procedure: Quadratus Lumborum Block — Quadratus Lumborum Block will be performed using 0.25-0.5% cc/kg bupivacaine
  Arms: GROUP USING Quadratus Lumborum Block

SUMMARY:
Analgesia methods such as systemic analgesics, quadratus lumborum block, and transversus abdominis plane block are used for pain management after lower abdominal surgery. Quadratus lumborum block (QLB) requires the patient to be in the lateral decubitus position, and the drug injection point is deeper. Transversus abdominis plane (TAP) block, on the other hand, can be performed with the patient supine, and the drug injection point is more superficial. However, while TAP block has no effect on visceral pain, QLB is also effective in visceral pain. Furthermore, although the injection point for QLB is deep, systemic absorption of the drug is expected to be lower than with TAP block due to its distance from vascular structures. Consequently, blood local anesthetic concentrations and the risk of local anesthetic systemic toxicity (LAST) are also expected to be lower. Despite the deeper injection, it is expected to provide better analgesia and a lower risk of LAST, making it superior to TAP block. This study aimed to compare the postoperative pain relief effect of quadratus lumborum block and transversus abdominis plane block, routinely performed in the clinic to prevent postoperative pain in pediatric patients undergoing inguinal hernia surgery, using the FLACC (Face, Leg Mobility, Activity, Crying, and Consolability) score for blood bupivacaine dose after drug injection. Based on these data, if lower blood drug concentrations are detected in patients undergoing QLB, the investigators aim to implement this technique routinely in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective inguinal hernia surgery.
* 1-6 years of age
* ASA I-II patients

Exclusion Criteria:

* Vulnerable populations such as those incapacitated, those in intensive care, those unconscious, those unable to give personal consent, or impressionable individuals will not be included in the study.
* Although pediatric patients who may be considered a vulnerable population will be included in the study, patients with serious illnesses such as ASA III-IV will not be included in this group.
* Patients who refuse to participate in the observational study, their parents/legal guardians,
* Patients with incomplete data
* Patients who underwent surgery with an incision other than the planned one for any reason.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Blood bupivacaine level | 30 and 60 minutes after block application
  After the block application, 2 mL of blood will be taken into a routine biochemistry tube and the blood bupivacaine level will be measured.
FLACC (Face, Leg Mobility, Activity, Crying, Consolation) | 0.HOUR, 1.HOUR, 2.HOUR, 4.HOUR, 6.HOUR, 12.HOUR 24.HOUR
  To compare postoperative pain efficacy with FLACC (Face, Leg Mobility, Activity, Crying, Consolability) Minimum score is 0 (no pain), maximum score 10 (the worse pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided